CLINICAL TRIAL: NCT05009472
Title: Evaluation of the Treatment Outcome of Cleft Palate Patients Treated With Differential Opening Expander With Rapid Protocol and Face Mask Using CBCT
Brief Title: Rapid Maxillary Expansion and Protraction by Expander Differential Opening EDO in Cleft Lip and Palate Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Taghreed riyadh saleh alazzawi, principal investigator, Faculty of Dental Medicine for Girls
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORTHO-109-2-E
Record Dates: First submitted 2021-07-29; First posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Cleft Lip and Palate
Keywords: cleft palate patient; Rapid maxillary expansion RME; cone beam computed tomography CBCT; expansion; face mask
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cleft Lip and Palate Patient (Experimental): Cleft patient with transverse maxillary constriction and anteroposterior deficiency
  Interventions: Device: expander with deferential opening and petit face mask

INTERVENTIONS:
Device: expander with deferential opening and petit face mask — bonded expander with two screws and vertical hooks for attachment face mask. adjustment face mask with forehead and chin anchorage

SUMMARY:
maxillary expansion in cleft palate patient with expander and using face mask.

DETAILED DESCRIPTION:
patient with cleft palate and maxillary constriction, deficiency will be treat using expander with differential opening which has two screws on anteriorly and another posteriorly positional in midline palate anteriorly as much as possible.

rapid maxillary expansion will be using one turns in day(two turns in the morning and two turns in the evening).

with petit face mask for maxillary protraction and superimposition CBCT will be taken between before and after treatment .

ELIGIBILITY:
Inclusion Criteria:

* ● Patients of both sexes.

  * Cleft lip and palate patients.
  * All patient age range 8-12 years.
  * All the case showed maxillary arch constriction and deficiency.
  * All patients had maxillary permanent first molars.
  * Primary lip adhesion and palatal closure.

Exclusion Criteria:

* • Absent maxillary permanent first molars.

  * Patients had received any surgical assisted rapid maxillary expansion, maxillary protraction or fixed orthodontics before.
  * Less than two dental unit beside maxillary first molar.
  * Uncooperative patients/parents.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2021-06-26 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Changes in 3 dimensions of skull before and after expansion | Six months
  Full skull Cone Beam Computerized Tomography

CONTACTS AND LOCATIONS:
Overall Officials: dr. mohsena ahmad, phd, Study Director — Lecturer of orthodontics department Faculty of Dental Medicine for Girls Alazhar univercity
Locations (2):
- Egypt (2):
  - Faculty of Dental Medicine for Girls Al-Azhar University, Cairo, Nasr City
  - Taghreddd, Cairo

IPD SHARING:
Plan to Share IPD: No
treatment cleft lip and palate patient with EDO with rapid protocol and face mask

REFERENCES:
- See also: Rapid maxillary expansion and face mask with class III malocclusion — http://doi.org/10.2319/092913-707.1